CLINICAL TRIAL: NCT05305092
Title: Integrated PET/MRI Study of Cognitive Impairment in Premenopausal Breast Cancer Patients After Chemotherapy or Endocrine Therapy
Brief Title: Assessment of Brain Cognitive Impairment in Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Collaborators: Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 82071993
Record Dates: First submitted 2022-03-06; First posted 2022-03-31 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Chemo-brain; Endocrine Therapy
Keywords: CRCI; psycho-behavioral technology; Integrated PET/MRI technology; Biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, gut microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chemotherapy: Premenopausal breast cancer patients receiving chemotherapy (including preoperative neoadjuvant chemotherapy) and endocrine therapy after surgery
  Interventions: Device: PET/MRI, psychobehavioral tests and questionnaires, serum biomarkers and stool sample
- Endocrine therapy: Premenopausal breast cancer patients receiving endocrine therapy alone after surgery
  Interventions: Device: PET/MRI, psychobehavioral tests and questionnaires, serum biomarkers and stool sample
- Healthy control: Healthy non-cancer controls
  Interventions: Device: PET/MRI, psychobehavioral tests and questionnaires, serum biomarkers and stool sample

INTERVENTIONS:
Device: PET/MRI, psychobehavioral tests and questionnaires, serum biomarkers and stool sample — Neuroimaging data were collected by integrated PET/MRI machine, and collected the psychobehavioral data, the serum and stool samples of participants.

SUMMARY:
To explore the cognitive impairment caused by chemotherapy and endocrine therapy in premenopausal breast cancer patients and to find biomarkers with early predictive effect on this cognitive impairment by using multimodal integrated PET/MRI technology combined with psychobehavioral technology.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women worldwide, and cancer-related cognitive impairment (CRCI) has become one of the most concerning clinical problems in breast cancer treatment. This project intends to use the combination of advanced PET/MRI technology and psycho-behavioral methods to observe the cognitive impairment and the changes in brain structure, function and glucose metabolism caused by chemotherapy and endocrine therapy in premenopausal breast cancer patients, then looking for possible predictors, through early identification of patients at risk of cognitive decline after chemotherapy or endocrine therapy, to provide a scientific basis for the rational selection of breast cancer treatment plans in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary stage I-II breast cancer.
* Premenopausal women (menopausal status determined by National Comprehensive Cancer Network Breast Cancer Guidelines criteria).
* No treatment other than surgery has been started (if neoadjuvant chemotherapy is required before surgery, enroll before chemotherapy starts).
* Eastern Cooperative Oncology Group score of 0-1 points.
* Can understand and complete various scales.
* Right handedness.
* Female subjects of childbearing potential must be willing to use a medically-approved high-efficiency contraceptive method (eg, intra-uterine device, birth control pill, or condom) for the duration of the study.
* Sign the informed consent and voluntarily participate in this clinical observation.

Exclusion Criteria:

* Central nervous system (CNS) disease, history of malignancy, chronic loss of consciousness, head trauma, and any disease affecting cognitive function.
* Current or former epilepsy, dementia, or learning disabilities.
* Past psychiatric history.
* Past history of malignancy.
* MRI related contraindications: pacemakers, defibrillators, hearing aids, insulin pumps, drug dose control devices and other metal implants; patients with severe hyperthermia; patients with claustrophobia.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Premenopausal patients with stage I-II breast cancer.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change of gray matter volume of whole brain | Baseline, 6,18,30 months later
  Gray matter volume will be measured with magnetic resonance imaging (high resolution T1-weighted image)
Change of white matter integrity of whole brain. | Baseline, 6,18,30 months later
  Fractional anisotropy, axial diffusivity and radial diffusivity will be measured with magnetic resonance imaging (diffusion tensor imaging)
Change of metabolism of glucose in the brain | Baseline, 6,18,30 months later
  Accumulation of 18F-fluorodeoxyglucose(18F-FDG) will be analyzed by time-related Positron emission tomography
Change of functional connectivity of whole brain | Baseline, 6,18,30 months later
  Functional connectivity will be measured with magnetic resonance imaging based on blood oxygen level dependence
Change of verbal learning and memory | Baseline, 6,18,30 months later
  Verbal learning and memory scores will be assessed with Hopkins Verbal Learning Test-Revised.The minimum value is 0, and the maximum value is 12. The higher scores mean a better outcome.
Change of information processing speed | Baseline, 6,18,30 months later
  Information processing speed scores will be assessed with Wechsler Adult Intelligence Scale(WAIS-III) Digit Symbol Coding score.The minimum value is 0, and the maximum value is 90. The higher scores mean a better outcome.
Change of executive function | Baseline, 6,18,30 months later
  Executive function scores will be assessed with Stroop color-word test.The minimum value is 0, and the maximum value is 50. The higher scores mean a better outcome.
Change of attention, verbal short term and working memory | Baseline, 6,18,30 months later
  Attention, verbal short term and working memory scores will be assessed with Digit span.The minimum value is 0, and the maximum value is 12. The higher scores mean a better outcome.
Change of life quality. | Baseline, 6,18,30 months later
  Quality of life scores will be assessed with Quality-of-Life Questionnaire C30. The minimum value is 30, and the maximum value is 126. The higher scores mean a worse outcome.
Change of anxiety | Baseline, 6,18,30 months later
  Anxiety scores will be assessed with Self-Rating Anxiety Scale.The minimum value is 20, and the maximum value is 80. The higher scores mean a worse outcome.
Change of depression | Baseline, 6,18,30 months later
  Depression scores will be assessed with Self-rating depression scale.The minimum value is 20, and the maximum value is 80. The higher scores mean a worse outcome.
Change of fatigue | Baseline, 6,18,30 months later
  Fatigue scores will be assessed with Fatigue Severity Scale. The minimum value is 9, and the maximum value is 63. The higher scores mean a worse outcome.
Change of sleep | Baseline, 6,18,30 months later
  Sleep scores will be assessed with Pittsburgh sleep quality index.The minimum value is 9, and the maximum value is 36. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of the concentration of serum biomarkers. | Baseline, 6,18,30 months later
  The concentration of GFAP with pg/mL, S-100B with pg/mL，IL-6 with pg/mL, IL-8 with pg/mL, IL-10 with pg/mL, IL-1β with pg/mL, TNF-α with pg/mL, UCH-L1 with pg/mL, NSE with pg/mL, T-Tau with pg/mL, P-Tau with pg/mL, NFL with pg/mL, BDNF with pg/mL, and VEGF with pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Menghui Yuan, phd, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China